CLINICAL TRIAL: NCT00737880
Title: A Prospective Randomized Multicenter Trial Comparing Histidine-Tryptophane-Ketoglutarate (HTK) Versus University of Wisconsin (UW) Perfusion Solution in Clinical Pancreas Transplantation
Brief Title: Histidine-Tryptophane-Ketoglutarate (HTK) vs University of Wisconsin (UW) Perfusion in Clinical Pancreas Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: University Hospital, Ghent (Other); University of Rostock (Other); Charite University, Berlin, Germany (Other); Dr. F. Köhler Chemie GmbH (Industry)
Responsible Party: Prof. Dr. Alfred Königsrainer, Transplantation Surgery / Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-KSM-III/6/00
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Diabetes Mellitus; Pancreas Transplantation
Keywords: Pancreas Clinical, Donor; Pancreas Clinical, Preservation Solutions; Organ Preservation and Procurement, Surgery; Organ Procurement, Ischemia reperfusion Injury; Organ Preservation and Procurement
MeSH Terms: conditions — Diabetes Mellitus; Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): In situ organ perfusion using HTK solution during pancreas procurement
  Interventions: Other: Organ perfusion during pancreas procurement
- 2 (Active Comparator): In situ perfusion using UW solution during pancreas procurement
  Interventions: Other: Organ perfusion during pancreas procurement

INTERVENTIONS:
Other: Organ perfusion during pancreas procurement — Usage of UW or HTK perfusion solution during in situ abdominal organ perfusion in multi-organ procurement

SUMMARY:
Graft preservation in clinical pancreas transplantation is based on hypothermia achieved by topic cooling and cold in situ flushing using special perfusion solutions designed to attenuate the effects of ischemia/reperfusion and prolong cold ischemia tolerance.

For pancreas transplantation, University of Wisconsin (UW) solution is the most commonly used perfusate. However, over the last years, Histidine-Tryptophan-Ketoglutarate (HTK) solution has been increasingly used for abdominal organ procurement. Retrospective reports published so far have demonstrated the safety of both perfusion solutions.

However, to date, no prospective study comparing both perfusion solutions has been published. Aim of this study was to prospectively evaluate early pancreas graft function in clinical pancreas transplantation after organ perfusion with HTK vs. UW solution.

The study hypothesis is that HTK is not inferior to UW for organ perfusion during procurement in clinical pancreas transplantation.

ELIGIBILITY:
Inclusion Criteria:

* brain dead, heart beating organ donor
* donor age 10 - 50 years
* donor body mass index < 30kg/m2
* pancreas cold ischemia time < 20 hours
* written informed consent of the pancreas recipient

Exclusion Criteria:

* missing written consent
* pancreas retransplantation
* recipient participation in another study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2001-07; Primary Completion 2004-01 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Pancreas graft survival | 6 months after transplantation

SECONDARY OUTCOMES:
Serum amylase | 6 months after transplantation
Serum lipase | 6 months after transplantation
C-peptide | 6 months after transplantation
HbA1c | 6 months after transplantation
Exogenous insulin requirement | 6 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Königsrainer, Prof., M.D., Principal Investigator — Transplantat Surgery, Medical University Innsbruck
Locations (4):
- Center of Operative Medicine / Department of Visceral, Transplant and Thoracic Surgery / Medical University Innsbruck, Innsbruck, Tyrol, Austria
- Department of General, Hepato-Biliary and Transplantation Surgery, Ghent, Belgium
- Germany (2):
  - Department of General, Visceral and Transplantation Surgery, Charite Campus Virchow Klinikum, Humboldt University Berlin, Berlin, State of Berlin
  - Department of General, Vascular, Thoracic and Transplantation Surgery, University of Rostock, Rostock

REFERENCES:
- [Derived] Schneeberger S, Biebl M, Steurer W, Hesse UJ, Troisi R, Langrehr JM, Schareck W, Mark W, Margreiter R, Konigsrainer A. A prospective randomized multicenter trial comparing histidine-tryptophane-ketoglutarate versus University of Wisconsin perfusion solution in clinical pancreas transplantation. Transpl Int. 2009 Feb;22(2):217-24. doi: 10.1111/j.1432-2277.2008.00773.x. Epub 2008 Oct 24. PMID 18954363